CLINICAL TRIAL: NCT03750266
Title: The Role of 3D Images and Models to Aid Management of Cases of Congenital Diaphragmatic Hernia Diagnosed in the Antenatal Period. Consecutive Patients Studied From Diagnosis to Post Operative Period.
Brief Title: 3D Animation and Models to Aid Management of Fetal CDH
Status: Recruiting | Type: Observational
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH19783
Record Dates: First submitted 2018-08-14; First posted 2018-11-23 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital Diaphragmatic Hernia referred for fetal MRA
  Interventions: Other: No intervention data collected through routine scans

INTERVENTIONS:
Other: No intervention data collected through routine scans — No intervention, we wish to use the images a mother would have done as part of her normal medical care and make both 3D animations and 3D models of the baby and it's CDH.

SUMMARY:
We wish to use the images a mother would have done as part of her normal medical care and make both 3D animations and 3D models of the baby and it's CDH. This will both help the parents see what the problem is and also allow the surgeons, who will operate on the baby once it has been born, to see the size of the hole and what organs are in the wrong place.

ELIGIBILITY:
Inclusion Criteria:

* Target Population: pregnancy women attending Jessop Wing Fetal medicine unit.
* Accessible population: Pregnant women attending Jessop Wing Fetal medicine unit. Whose fetus had a CDH and are referred to MRI.
* Study population: Pregnant women attending Jessop Wing Fetal medicine unit. Whose fetus had a CDH and are referred to MRI and agree to take part in the study.

Exclusion Criteria:

* Not able to give informed consent due to any reason including poor understanding of English
* Under 18 years of age.
* Unable to complete the fetal MRI process due to either metal implants or claustrophobia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women whose fetus had a CDH and are referred to MRI.
Study Population: Pregnant women attending Jessop Wing Fetal medicine unit. Whose fetus had a CDH and are referred to MRI and agree to take part in the study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-10-04 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Patient demographics | Baseline
  Gestational age at time of scan and health outcomes from patient notes. This will be used to assess the accuracy of the 3D models developed.

CONTACTS AND LOCATIONS:
Locations (1):
- Jessop Wing Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No